CLINICAL TRIAL: NCT02187783
Title: Modular Phase II Study to Link Targeted Therapy to Patients With Pathway Activated Tumors: Module 8 - LEE011 for Patients With CDK4/6 Pathway Activated Tumors
Brief Title: LEE011 for Patients With CDK4/6 Pathway Activated Tumors (SIGNATURE)
Acronym: SIGNATURE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLEE011XUS03
Record Dates: First submitted 2014-07-09; First posted 2014-07-11 (Estimated); Results first posted 2019-04-16 (Actual); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: Tumors With CDK4/6 Pathway Activation
Keywords: Solid malignancy; Hematologic malignancy; Mutations; Amplifications; Signature; CDK4; CDK6; CDK4/6; Cyclin D1; CCND,; Cyclin D3; p16 mutation; CDKN2A; LEE011; Breast cancer; Ovarian cancer; Lymphoma; Mesothelioma; Pancreatic neuroendocrine; Leukemia; Tumor
MeSH Terms: conditions — Hematologic Neoplasms; Breast Neoplasms; Ovarian Neoplasms; Lymphoma; Mesothelioma; Leukemia; Neoplasms | interventions — ribociclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- LEE011 (Experimental): LEE011 600 mg (hard gelatin capsules) was administered orally once daily for 3 weeks on/1 week off. A complete treatment cycle was defined as 28 days.
  Interventions: Drug: LEE011

INTERVENTIONS:
Drug: LEE011 — Study drug was provided in 200 mg and 50 mg hard gelatin capsules to be taken orally

SUMMARY:
The purpose of this signal seeking study was to determine whether treatment with LEE011 demonstrates sufficient efficacy in CDK4/6 pathway activated solid tumors and/or hematologic malignancies to warrant further study.

ELIGIBILITY:
Inclusion Criteria:

* Patient had a confirmed diagnosis of a select solid tumor (except breast cancer (however, triple negative was included), liposarcoma, CRPC, melanoma and teratoma) or hematological malignancy (except mantle cell lymphoma).
* Patient must have been pre-identified as having a tumor with CDK4 amplification or mutation, CDK6 amplification or mutation, Cyclin D1 (CCND1) amplification, Cyclin D3 (CCND3) amplification, or p16 (CDKN2A) mutation
* Patient had received at least one prior treatment for recurrent, metastatic and /or locally advanced disease and for whom no standard therapy options are anticipated to result in a durable remission.
* Patient had progressive and measurable disease as per RECIST 1.1. or other appropriate hematological guidelines.
* Patient had an Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1

Exclusion Criteria:

* Patients had received prior treatment with LEE011.
* Patient had clinically significant resting bradycardia (heart rate < 50 at rest), tachycardia (heart rate > 90 at rest), PR interval > 220 msec, QRS interval > 109 msec, or QTcF > 450 msec.
* Patients had primary CNS tumor or CNS tumor involvement
* Patient had received chemotherapy or anticancer therapy ≤ 4 weeks prior to starting study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2014-08-25 (Actual); Primary Completion 2018-01-17 (Actual); Study Completion 2018-01-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (61):
- United States (61):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Alaska Clinical Research, Anchorage, Alaska
  - Arizona Oncology Associates Dept. Of Onc., Phoenix, Arizona
  - University of Arkansas/ Arkansas Cancer Research Center UA Medical Sciences, Little Rock, Arkansas
  - PCR Oncology, Pismo Beach, California
  - University of California Davis Cancer Center UC Davis Cancer (3), Sacramento, California
  - Sarah Cannon Research Institute, Denver, Colorado
  - Danbury Hospital, Danbury, Connecticut
  - Yale University School of Medicine Smilow Cancer Hospital, New Haven, Connecticut
  - Whittingham Cancer Center Norwalk Hospital, Norwalk, Connecticut
  - Stamford Hospital Med. Oncology Hematology Res., Stamford, Connecticut
  - Florida Hospital Cancer Institute, Orlando, Florida
  - NorthWest Georgia Oncology Centers NW Georgia Oncology, Marietta, Georgia
  - Harbin Clinic Medical Oncology Clin. Res., Rome, Georgia
  - Queen's Medical Center Queens Cancer Center, Honolulu, Hawaii
  - Northwestern Medicine Developmental Therapeutics Institute, Chicago, Illinois
  - Indiana University Indiana Univ. - Purdue Univ., Indianapolis, Indiana
  - Northern Indiana Cancer Research Consortium No. Indiana Cancer Res., South Bend, Indiana
  - University of Iowa Hospitals & Clinics Regulatory Contact 2, Iowa City, Iowa
  - New England Cancer Specialists, Scarborough, Maine
  - St. Agnes Hospital St. Agnes Hospital (2), Baltimore, Maryland
  - Michigan Medicine University of Michigan Int. Medicine Oncology, Ann Arbor, Michigan
  - Cancer and Hematology Centers of West Michigan Dept. of Oncology, Grand Rapids, Michigan
  - Saint Luke's Hospital/Marion Bloch Neuroscience Institute St. Luke's Hospital (4), Kansas City, Missouri
  - Research Medical Center Research Med Center (2), Kansas City, Missouri
  - Comprehensive Cancer Centers of Nevada CCC of Nevada- Southwest (2), Las Vegas, Nevada
  - Cooper Health System Cooper Health System (5), Camden, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - New Mexico Cancer Care Alliance, Albuquerque, New Mexico
  - Cancer Center at Presbyterian, Albuquerque, New Mexico
  - Broome Oncology Broome Oncology (2), Johnson City, New York
  - University of N C at Chapel Hill Physician Office Building, Chapel Hill, North Carolina
  - Carolina Oncology Specialists, PC, Hickory, North Carolina
  - Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Oncology Hematology Care Inc Oncology Hematology Care 2, Cincinnati, Ohio
  - Cleveland Clinic Foundation Taussig Cancer Institute, Cleveland, Ohio
  - Ohio State University Medical Center Comprehensive Cancer Center, Columbus, Ohio
  - Oregon Health and Science University Oregon Health & Science U (56), Portland, Oregon
  - Salem Health, Salem, Oregon
  - Fox Chase Cancer Center Dept of Medical Oncology, Philadelphia, Pennsylvania
  - Rhode Island Hospital Rhode Island Hosp. (2), Providence, Rhode Island
  - Greenville Health System ITOR - Cancer Institute, Greenville, South Carolina
  - Sanford University of South Dakota Medical Center Sanford Health, Sioux Falls, South Dakota
  - Chattanooga Oncology and Hematology Assoicates, PC Chattanooga Oncology, Chattanooga, Tennessee
  - The West Clinic Dept. of the West Clinic, Memphis, Tennessee
  - Tennessee Oncology Tennessee Oncology (3), Nashville, Tennessee
  - Coastal Bend Cancer Center, Corpus Christi, Texas
  - Oncology Consultants Oncology Group, Houston, Texas
  - MD Anderson Cancer Center/University of Texas MD Anderson Cancer Center (3), Houston, Texas
  - University of Texas Health Science Center at San Antonio Cancer Therapy & Research Ctr., San Antonio, Texas
  - Intermountain Medical Center Intermountain Healthcare, Murray, Utah
  - Utah Cancer Specialists Utah Cancer Specialists (11), Salt Lake City, Utah
  - Shenandoah Oncology Shenadoah Oncology (2), Winchester, Virginia
  - Kadlec Clinic Hematology and Oncology Kadlec Clinic Hematology & Onc, Kennewick, Washington
  - Vista Oncology Inc. PS, Olympia, Washington
  - Multicare Research Institute, Tacoma, Washington
  - Northwest Medical Specialties Rainier Physicians, PC, Tacoma, Washington
  - Providence St. Mary Regional Cancer Center, Walla Walla, Washington
  - Wenatchee Valley Medical Center Wenatchee Valley, Wenatchee, Washington
  - Aurora Research Institute Aurora Health Care, Milwaukee, Wisconsin
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There were 176 patients screened
Groups:
- Ribociclib 600 mg: LEE011 600 mg (hard gelatin capsules) was administered orally once daily for 3 weeks on/1 week off. A complete treatment cycle was defined as 28 days.
Period: Overall Study
Arm/Group | Ribociclib 600 mg
Started | 106
Patients With Solid Tumors | 105
Completed | 0
Not Completed | 106
Not completed — Adverse Event | 8
Not completed — Death | 3
Not completed — Progressive disease | 80
Not completed — Protocol Violation | 3
Not completed — Physician Decision | 2
Not completed — Withdrawal by Subject | 9
Not completed — Study terminated by sponsor | 1

BASELINE CHARACTERISTICS:
Arm/Group | Ribociclib 600 mg
Number analyzed (Participants) | 106
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.5 (13.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56
  Male | 50
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 90
  Black or African American | 4
  Asian | 5
  Other | 7
Primary tumor type [Count of Participants; unit: Participants] — Primary tumor type was sponsor adjudicated.
  Participants
    Adrenals | 1
    Bladder | 7
    Breast-triple negative | 7
    Cervix | 1
    Cholangio | 2
    Chordoma | 1
    Colorectal | 2
    Esophagus | 3
    Gall bladder ducts | 1
    Gastroesophageal junction | 4
    Gastrointestinal stromal tumor | 1
    Head and neck non-squamous cell carcinoma | 4
    Head and neck squamous cell carcinoma | 7
    Kidneys | 2
    Liver | 2
    Lung non-small cell adenocarcinoma | 9
    Lung non-small cell non-adenocarcinoma | 2
    Lung non-small cell squamous | 6
    Lymphoma | 1
    Mesothelioma | 5
    Neuroendocrine | 2
    Ovarian | 3
    Pancreas | 5
    Penile | 1
    Prostate | 1
    Salivary gland | 1
    Sarcoma | 13
    Skin non-melanoma | 3
    Thyroid | 1
    Unknown primary | 4
    Uterus | 4
Number of participants who had radiotherapy, surgery and liver metastasis [Count of Participants; unit: Participants]
  Prior antineoplastic radiotherapy | 61
  Prior antineoplastic surgery | 92
  Liver metastasis | 29
Eastern Cooperative Oncology Group (ECOG) Performance Status for participants [Number; unit: participants] — ECOG: 0 = Fully active, able to carry on all pre-disease performance without restriction; 1 = Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g. light housework, office work; 2 = Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours; 3 = Capable of only limited self-care, confined to bed or chair more than 50% of waking hours; 4 = Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair; 5 = Dead.
  participants
    Performance status = 0 | 36
    Performance status = 1 | 70

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Solid Tumor Response ≥ 16 Weeks for Based Upon Local Investigator Assessments
Description: Clinical benefit (CB) for patients with solid tumors were assessed using RECIST 1.1 and included responses of Complete Response (CR) or Partial Response (PR) or Stable Disease (SD) for ≥ 16 weeks. CR and PR (for solid tumors) required a confirmation at least 4 weeks after the initial response observation. For hematologic tumors other appropriate hematological response criteria was applied. CR=Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have had reduction in short axis to <10 mm, PR=At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters, SD=Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study, PD=At least a 20% increase in the sum of diameter of all measured target lesions and also demonstrate an absolute increase of at least 5 mm. FAS
Time Frame: Baseline up ≥16 weeks up to approximately 36 months
Measure: Count of Participants; unit: Participants
Arm/Group | Ribociclib 600 mg
Number analyzed (Participants) | 105
Participants
  Complete response | 0
  Partial response (PR) | 3
  Stable disease (SD) | 16
  Progressive disease (PD) | 71
  Non-evaluable (NE) | 15

2. Primary Outcome: Clinical Benefit Rate (CBR) of ≥ 16 Weeks FAS
Description: CBR was determined by local, Investigator assessment for each tumor assessment and defined as responses of CR + PR + SD for ≥ 16 weeks. CR and PR (for solid tumors) required a confirmation at least 4 weeks after the initial response observation. For hematologic tumors other appropriate hematological response criteria was applied. CR=Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have had reduction in short axis to <10 mm, PR=At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters, SD=Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study, PD=At least a 20% increase in the sum of diameter of all measured target lesions and also demonstrate an absolute increase of at least 5 mm FAS
Time Frame: Baseline and ≥ 16 weeks up to approximately 36 months
Measure: Number (95% Confidence Interval); unit: participant
Arm/Group | Ribociclib 600 mg
Number analyzed (Participants) | 105
participant | 19 [11.3 to 26.8]

3. Secondary Outcome: Progression Free Survival (PFS)
Description: Progression-free survival (PFS) is the time from the date of start of treatment to the date of event defined as the first documented progression or death due to any cause within 30 days of the last dose. If a subject has not had an event, progression-free survival is censored at the date of last adequate tumor assessment. Progressive disease is defined as at least a 20% increase in the sum of diameter of all measured target lesions, taking as reference the smallest sum of diameter of all target lesions recorded at or after baseline. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm (Note: the appearance of one or more new lesions is also considered progression)
Time Frame: Every 8 weeks until death, assessed up to 24 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ribociclib 600 mg
Number analyzed (Participants) | 106
months | 1.8 [1.8 to 1.9]

4. Secondary Outcome: Overall Survival (OS)
Description: Number of participants Overall survival (OS) is defined as the time from the date of first dose to the date of death due to any cause.
Time Frame: Baseline up to approximately 36 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ribociclib 600 mg
Number analyzed (Participants) | 106
months | 7.7 [5.3 to 9.2]

5. Secondary Outcome: Number of Days for Duration of Response for Responders
Description: Duration of response (DOR) is defined as time from the first documented response to the date first documented disease progression or relapse or death due to any cause. For patients with solid tumors the assessment criteria will be RECIST 1.1 and will include responses of CR and/or PR.
Time Frame: Baseline up to approximately 36 months
Measure: Number; unit: Days
Arm/Group | Ribociclib 600 mg
Number analyzed (Participants) | 3
Days
  Patient 1 | 254
  Patient 2 | 330
  Patient 3 | 985

6. Primary Outcome: Overall Response Rate (ORR) ≥ 16 Weeks. FAS
Description: ORR was determined by local, Investigator assessment for each tumor assessment and defined as responses of CR+PR ≥ 16 weeks. FAS
Time Frame: Baseline and ≥ 16 weeks up to approximately 36 months
Measure: Number (95% Confidence Interval); unit: participant
Arm/Group | Ribociclib 600 mg
Number analyzed (Participants) | 105
participant | 3 [0.6 to 8.1]

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected from First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV). All AEs reported in this record are from date of First Patient First Treatment until Last Patient Last Visit) which was an average of 2.7 months up to maximum of 36.2 months.
Arm/Group | Ribociclib 600 mg
All-Cause Mortality (participants affected / at risk) | 14/106
Serious Adverse Events (participants affected / at risk) | 40/106
Other Adverse Events (participants affected / at risk) | 104/106
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ribociclib 600 mg (N=106)
Anaemia (Blood and lymphatic system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Cardio-respiratory arrest (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 1
Pericardial effusion (Cardiac disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 2
Abdominal pain upper (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 1
Mouth haemorrhage (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 3
Small intestinal obstruction (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 2
Non-cardiac chest pain (General disorders) | 1
Pain (General disorders) | 2
Abscess (Infections and infestations) | 1
Peritonitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Pseudomonal sepsis (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 1
Pyelonephritis acute (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Blood bilirubin increased (Investigations) | 1
Weight decreased (Investigations) | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1
Failure to thrive (Metabolism and nutrition disorders) | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 1
Malnutrition (Metabolism and nutrition disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Aphasia (Nervous system disorders) | 1
Embolic stroke (Nervous system disorders) | 1
Transient ischaemic attack (Nervous system disorders) | 1
Confusional state (Psychiatric disorders) | 1
Mental status changes (Psychiatric disorders) | 1
Nephropathy toxic (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Renal tubular necrosis (Renal and urinary disorders) | 1
Ureteric obstruction (Renal and urinary disorders) | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2
Deep vein thrombosis (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
Thrombophlebitis superficial (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ribociclib 600 mg (N=106)
Anaemia (Blood and lymphatic system disorders) | 26
Leukopenia (Blood and lymphatic system disorders) | 12
Neutropenia (Blood and lymphatic system disorders) | 33
Thrombocytopenia (Blood and lymphatic system disorders) | 13
Abdominal pain (Gastrointestinal disorders) | 10
Constipation (Gastrointestinal disorders) | 21
Diarrhoea (Gastrointestinal disorders) | 28
Dyspepsia (Gastrointestinal disorders) | 8
Nausea (Gastrointestinal disorders) | 46
Vomiting (Gastrointestinal disorders) | 31
Asthenia (General disorders) | 8
Chest pain (General disorders) | 8
Fatigue (General disorders) | 45
Oedema peripheral (General disorders) | 12
Pyrexia (General disorders) | 8
Urinary tract infection (Infections and infestations) | 11
Alanine aminotransferase increased (Investigations) | 11
Aspartate aminotransferase increased (Investigations) | 11
Blood alkaline phosphatase increased (Investigations) | 8
Blood creatinine increased (Investigations) | 15
Electrocardiogram QT prolonged (Investigations) | 12
Gamma-glutamyltransferase increased (Investigations) | 9
Lymphocyte count decreased (Investigations) | 8
Neutrophil count decreased (Investigations) | 16
Platelet count decreased (Investigations) | 9
Weight decreased (Investigations) | 9
White blood cell count decreased (Investigations) | 19
Decreased appetite (Metabolism and nutrition disorders) | 21
Dehydration (Metabolism and nutrition disorders) | 7
Hyperglycaemia (Metabolism and nutrition disorders) | 9
Hypoalbuminaemia (Metabolism and nutrition disorders) | 7
Hypokalaemia (Metabolism and nutrition disorders) | 7
Hypomagnesaemia (Metabolism and nutrition disorders) | 9
Arthralgia (Musculoskeletal and connective tissue disorders) | 8
Back pain (Musculoskeletal and connective tissue disorders) | 12
Muscular weakness (Musculoskeletal and connective tissue disorders) | 7
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 8
Myalgia (Musculoskeletal and connective tissue disorders) | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7
Dizziness (Nervous system disorders) | 13
Headache (Nervous system disorders) | 9
Anxiety (Psychiatric disorders) | 7
Confusional state (Psychiatric disorders) | 6
Insomnia (Psychiatric disorders) | 11
Proteinuria (Renal and urinary disorders) | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 15
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 20
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6
Rash (Skin and subcutaneous tissue disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Statistical Analysis Plan (2015-09-27): https://cdn.clinicaltrials.gov/large-docs/83/NCT02187783/SAP_000.pdf
  • Study Protocol (2017-04-10): https://cdn.clinicaltrials.gov/large-docs/83/NCT02187783/Prot_001.pdf